CLINICAL TRIAL: NCT04390217
Title: A Phase 2 Study to Evaluate LB1148 for the Treatment of Pulmonary Dysfunction Associated With COVID-19 Pneumonia
Brief Title: LB1148 for Pulmonary Dysfunction Associated With COVID-19 Pneumonia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company focused on other clinical programs
Sponsor: Leading BioSciences, Inc (Industry)
Responsible Party: Sponsor
Organization: Palisade Bio (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBS-COVID19-201
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Coronavirus Disease 2019; Covid19; COVID-19 Pneumonia
MeSH Terms: conditions — COVID-19 | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: All patients will be randomized into one of two treatment groups (LB1148 or Placebo) in a 1:1 ratio, and stratified by peripheral capillary oxygen saturation and by PF ratio at the time of Screening.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple blinding including the sponsor and all sponsor agents, subjects, investigators, care providers, and family members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LB1148 (Experimental): LB1148 contains 7.5 g TXA, polyethylene glycol (PEG), glucose, and electrolytes. A total of 700 mL of LB1148 Active will be administered daily as a split dose (350 mL, every 12 hours) for up to 7 days. LB1148 Active is given as a single bolus, to be delivered orally or enterally via NG/OG tube, and should be fully consumed or delivered within 2 hours of the start of administration.
  Interventions: Drug: LB1148
- Placebo (Placebo Comparator): Placebo contains polyethylene glycol (PEG), glucose, and electrolytes. A total of 700 mL of LB1148 Placebo will be administered daily as a split dose (350 mL, every 12 hours) for up to 7 days. LB1148 Placebo is given as a single bolus, to be delivered orally or enterally via NG/OG tube, and should be fully consumed or delivered within 2 hours of the start of administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB1148 — LB1148 is delivered orally/enterally, 700 mL per day split into two administrations of 350 mL, approximately 12 hours apart, for up to 7 days.
  Other Names: tranexamic acid (TXA)
  Arms: LB1148
Drug: Placebo — Placebo is delivered orally/enterally, 700 mL per day split into two administrations of 350 mL, approximately 12 hours apart, for up to 7 days.
  Arms: Placebo

SUMMARY:
This is a Phase 2, proof of concept, randomized, placebo-controlled, multicenter study to evaluate the ability of LB1148 to attenuate pulmonary dysfunction associated with COVID-19 pneumonia. The primary objective of this study is to determine if enteral administration of LB1148 will effect disease progression in hospitalized patients with moderate to severe COVID-19 via measurement of the proportion of subjects alive and free of respiratory failure at Day 28.

DETAILED DESCRIPTION:
The purpose of this study is to establish the safety and tolerability, along with preliminary evidence of efficacy, of LB1148 compared to placebo in hospitalized patients with moderate to severe coronavirus disease (COVID-19). All patients will be randomized into one of two treatment groups (LB1148 or Placebo) in a 1:1 ratio, and stratified by peripheral capillary oxygen saturation (SpO2) ≥ 93% on room air vs. < 93% on room air, and by PF ratio (PaO2, arterial oxygen partial pressure, to FiO2, fractional inspired oxygen) of ≥ 300 mmHg vs. PF ratio of < 300 mmHg at the time of Screening. (If PaO2 cannot be measured or acquired, SpO2 may be substituted to calculate the PF ratio.) LB1148 contains 7.5 g tranexamic acid (TXA), polyethylene glycol (PEG), glucose, and electrolytes. A total of 700 mL of LB1148 will be administered enterally, as a split dose (350 mL, every 12 hours). Study drug is given as a single bolus, to be delivered orally or via nasogastric (NG) or orogastric (OG) tube. For those patients assigned to placebo, a total of 700 mL of placebo will be administered enterally, as a split dose (350 mL, every 12 hours). The placebo contains PEG, glucose, and electrolytes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years of age or older) with the diagnosis of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, confirmed via an established standard reverse transcriptase polymerase chain reaction (RT-PCR) assay.
2. Patient or patient's legally authorized representative is willing and able to provide informed consent prior to performing any study-related procedures.
3. Patient is hospitalized and requires some form of supplemental oxygen, e.g., non-invasive ventilation, high flow oxygen device, or oxygen by mask or nasal cannula.
4. Patient has radiographic evidence of pulmonary infiltrate(s) or lung inflammation.

Exclusion Criteria:

1. Participation in any other interventional clinical trial using an experimental treatment (drug or device) for COVID-19.
2. Expected survival or time to withdrawal of life-sustaining treatments is expected to be < 7 days.
3. Patients with do not intubate orders.
4. Patients who require invasive mechanical ventilation at the time of Screening.
5. Patients who require renal replacement therapy (RRT) at the time of Screening.
6. Patients with known aspiration problems.
7. Has contraindications or potential risk factors to taking TXA. These include patients with:

   1. Known sensitivity to TXA;
   2. Recent craniotomy (past 30 days);
   3. Active cerebrovascular bleed;
   4. Active thromboembolic disease (such as deep vein thrombosis, pulmonary embolism, cerebral thrombosis, ischemic stroke, or acute coronary syndrome);
   5. Acute promyelocytic leukemia taking all-trans retinoic acid for remission induction
   6. Continuing use of a combined hormonal contraceptive and or combined hormonal replacement therapy (including combined hormonal pill, patch, or vaginal ring).
   7. Concomitant therapy with tissue plasminogen activators, Factor IX complex concentrates or anti-inhibitor coagulant concentrates.
8. Known medical history of congenital or acquired thrombophilia such as, but not limited to patients with:

   1. Sickle cell disease
   2. Nephrotic syndrome
   3. Factor V Leiden
   4. Prothrombin gene mutation
   5. Protein C or S deficiency
   6. Antithrombin III deficiency
   7. Antiphospholipid syndrome
9. Patients with myeloproliferative disorders.
10. Any other condition that, in the opinion of the treating Investigator, would preclude the patient from being an appropriate candidate for the study.
11. Female patients who are pregnant or breastfeeding at the time of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of LB1148 on disease progression via measurement of the proportion of patients who are alive and free of respiratory failure. | 28 Days
  The proportion of subjects alive and free of respiratory failure at Day 28.

SECONDARY OUTCOMES:
Clinical status at fixed time points | Measured at 3, 5, 7, 8, 10, 14 and 28 Days
  Number and proportion of patients with improved clinical status as assessed by a 9-point ordinal scale of disease severity at fixed timepoints (Days 3, 5, 7, 8, 10, 14, 28)
Duration of hospital stay | 28 Days
  Length of hospital stay (live discharge)
Measurement of the number and proportion of patients requiring admission to the intensive care unit (ICU) during hospitalization | 28 Days
  Number and proportion of patients requiring admission to the intensive care unit
Duration of ICU stay | 28 Days
  Length of ICU stay
Invasive mechanical ventilation requirements | 28 Days
  Number and proportion of patients requiring invasive mechanical ventilation
Duration of invasive mechanical ventilation | 28 Days
  Length of time patients require invasive mechanical ventilation
All-cause 28-day mortality | 28 Days
  The number and proportion of patients deceased at Day 28
Safety and tolerability of LB1148 | 28 Days
  The incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Dawson, MD, Study Director — Leading BioSciences, Inc

IPD SHARING:
Plan to Share IPD: No